CLINICAL TRIAL: NCT06260553
Title: Metronomic Oral Vinorelbine Combination With Tislelizumab in EGFR/ALK-negative Advanced NSCLC Patients Intolerant to First-line Standard Chemotherapy: A Singlearm Phase Il Clinical Trial
Brief Title: Metronomic Oral Vinorelbine Combination With Tislelizumab in EGFR/ALK-negative Advanced NSCLC
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOG008
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: EGFR/ ALK-negative Advanced NSCLC
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tislelizumab plus metronomic oral vinorelbine (Experimental)
  Interventions: Drug: tislelizumab and metronomic oral vinorelbine

INTERVENTIONS:
Drug: tislelizumab and metronomic oral vinorelbine — tislelizumab 200mg intravenous drip once every three weeks; Oral Vinorelbine 40mg three times a week for three weeks and Q28d for one course.

SUMMARY:
To evaluate the efficacy of metronomic chemotherapy combination with tislelizumab in EGFR/ALK-negative advanced NSCLC patients intolerant to first-line standard chemotherapy.

DETAILED DESCRIPTION:
This study is a clinical intervention study. The patients who comfirm the criteria will be treated with tislelizumab plus metronomic oral vinorelbine. The patients will be followed up until the tumor progressed, and the efficacy (PFS, ORR, DCR) of tumor therapy were evaluated. Drug administration regimen: tislelizumab 200mg intravenous drip once every 3 week3; Oral Vinorelbine 40mg three times a week for three weeks and Q28d for one course.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of stage IV (M1a or M1b-American Joint Committee on Cancer [AJCC] 8th edition) squamous NSCLC or non-squamous NSCLC without sensitising EGFR or ALK alterations.
* Has measurable disease based on RECIST 1.1 as determined by the local site investigator/radiology assessment.
* Has not received prior systemic treatment for metastatic NSCLC.
* Has a life expectancy of at least 3 months.
* Has fully understood this study and voluntarily signed a written informed consent form.
* Deemed unsuitable by the investigator for any platinum-doublet chemotherapy due to poor performance status (ECOG performance status of 2-3)；>= 75 years of age；substantial comorbidities; contraindication(s) for any platinum-doublet chemotherapy.

Exclusion Criteria:

* Histological or cytological confirmation of small cell lung cancer.
* Has a known history of prior malignancy except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has disorders of oral medication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-07 (Estimated); Primary Completion 2025-02-07 (Estimated); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  progression-free survival

SECONDARY OUTCOMES:
ORR | up to 12 months
  Objective Response Rate
DCR | up to 12 months
  Disease Control Rate
AE | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Number of Participants Who Experienced an Adverse Event

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No